CLINICAL TRIAL: NCT01743872
Title: Optical Imaging Measurement of Intravascular Solution Efficacy Trial
Acronym: OPTIMISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPTIMISE
Record Dates: First submitted 2012-09-26; First posted 2012-12-06 (Estimated); Results first posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-08

CONDITIONS: Peripheral Artery Disease
Keywords: Optical Coherence Tomography; Contrast; Dextran; Carbon Dioxide; Imaging; Catheter; Lower Extremity Artery
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Contrast Media; Dextrans

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- iOCT (Experimental): Arterial access will performed by the operating surgeon. An aortic and infrainguinal angiogram using the standard method of intravenous iodinated contrast under digital subtraction fluoroscopy will be conducted in the usual manner according to the vascular surgeon. A 54 mm section of Superficial Femoral Artery will be chosen for study imaging. An intervention sheath or injection catheter will be placed just proximal to the area of interest. An 0.014" wire will be passed distal to the area of interest. The patient will then undergo OCT of this 54mm section with each of the three mediums below using a continuous flushing method through injection catheter. All OCT imaging will be collected at a rate of 25mm/sec. In the event of a subsequent procedure, OCT imaging will again be performed
  Interventions: Procedure: Contrast Injection; Procedure: Dextran Injection; Procedure: CO2 Injection; Procedure: Heparinized Normal Saline Injection

INTERVENTIONS:
Procedure: Contrast Injection — Media #1: IV Contrast (Omnipaque 350) will be continuously injected at a rate range of 2.5-6ml/s for a maximum of 5 seconds. (Volume range of 12.5- 30ml) Intervention protocol will be followed per Cross-Reference Intervention.
Procedure: Dextran Injection — Media #2: Dextran 40 Solution will be continuously injected at a rate range of 2.5-6ml/s for a maximum of 5 seconds. (Volume range of 12.5- 30ml. Intervention protocol will be followed per Cross-Reference Intervention.
Procedure: CO2 Injection — Media #3: Carbon Dioxide (CO2) will be injected with large volume hand injection syringe as per the usual protocol. This be done with particular attention to avoid air in the closed system. In addition to supine, there is also an option that the patient's distal limb may be elevated to improve the flow of CO2 during injection. The surgeon will also wait at least 2 minutes between each CO2 injection to allow any potentially trapped CO2 to dissolve. A range of 20-60 ml will be used with each hand injection based on the data from the initial 5-10 pilot patients. Intervention protocol will be followed per Cross-Reference Intervention.
Procedure: Heparinized Normal Saline Injection — Media #4: Heparinized Normal Saline (Heparin NS) will be hand injected using 20 mL (2 U/mL) in antegrade fashion.

SUMMARY:
Iodinated contrast is the current gold standard for infrainguinal angiography imaging in patients without renal insufficiency and has also been used with intravascular Optical Coherence Tomography (iOCT) to improve image quality in human coronary arteries as well as carotid arteries. The current debate in the literature for iOCT medium is between iodinated contrast and dextran and CO2 may offer a superior method of iOCT imaging during lower extremity occlusive disease interventions.

The investigators hypothesize that the CO2 medium injection during iOCT data acquisition is feasible and will produce at least the same quality of imaging as that obtained with contrast or dextran without causing the problems of volume overload and renal toxicity seen with the two latter mediums.

Primary Outcomes Measured

* Quality: Cumulative number of clear image frame (CIF) through the entire 54mm length segment.
* Quantitative: Calculations of the area and diameter of each segment will be measured to determine if index of refraction has any effect between the three mediums to be tested.

The investigators expect to find little difference between all three iOCT mediums and hope to conclude that CO2 offers a superior side effect profile for iOCT imaging in the lower extremity arterial system.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) affects anywhere from 8-12 Million people in the United States. Many of these people go on to develop claudication, rest pain, and tissue loss. During the workup for these disease states many imaging modalities are conducted including Pulse Volume Recording, Duplex Ultrasound, Angiography, and IVUS, but an emerging catheter based imaging has been developed that may supplement the current modalities used.

Intravascular optical coherence tomography (iOCT) is based on near-infrared light system. The light reflects off plaque and other objects within vessels and the signals are processed into a series of axial images (A-scans) at different positions along the artery to generate a two-dimensional dataset (B-scans). These images are created at an extremely fine resolution of 10-15 μm, which has allowed iOCT to be used in many research settings including PAD and coronary artery disease. OCT has been approved for clinical use in the coronary territory by the FDA in May 2010. Since then many centers have been using iOCT in the daily clinical practice. However, it's still not widely in the clinical management of patients with PAD. There is hope that the high resolution capabilities of iOCT may help before and after an intervention to predict outcomes or correct errors in stent deployment.

The iOCT procedure for lower extremity PAD is fairly straightforward. An introducer is placed into the femoral artery. After which a wire is placed past the lesion of interest and the iOCT catheter is inserted. The catheter is then attached to an automated pullback device. Next an optical medium is needed to displace the erythrocytes. Due to the high resolution of the iOCT this is necessary for a cleaner image to analyze. At the time of injection of the optical medium a sensor triggers the catheter to be withdrawn (distal to proximal) at anywhere from 10-25 mm/sec. The images are captured and processed and arterial plaque can be characterized.

The greatest strength of the iOCT catheter is its high resolution images but the problem is that the imaging signal is substantially attenuated by blood. In order to remedy this complication techniques such as proximal balloon occlusion and continuous infusion of a fluid have been used to acquire improved iOCT images. In the continuous infusion methods, different mediums have been injected such as contrast, dextran, and even an oxygen-carrying substitute in hopes of improving decreasing the attenuation by blood.

In order the overcome the attenuation of red blood cells during iOCT imaging, we are proposing a novel approach involving CO2 injection to clear the erythrocytes. Currently CO2 is used as medium for digital subtraction angiography in patients with renal insufficiency and was first used in humans by Hawkins in 1982. The other alternative for angiography, iodinated contrast medium, is nephrotoxic and thus is avoided in these patients for fear of exacerbating the patient's acute or chronic problem. Another group where CO2 angiography is employed is history of a contrast allergy. Although this technique is usually used under these circumstances, Kerns et al reports conducting CO2 angiography in as high as 20% of their patients with abdominal and lower extremity studies.

In addition to the benefits of patients with allergies and renal insufficiency, CO2 is extremely safe in a variety of arterial and venous applications. It is 20 times as soluble as room air and is expired through the lungs in a first-pass-type effect. The current contraindication to CO2 digital subtraction angiography is that the cerebral arterial circulation should never be exposed to CO2 because of possible neurotoxicity. Relative contraindications include use in the presence of a large arteriovenous shunt, with nitrous oxide anesthesia, and used cautiously in patients with chronic obstructive pulmonary disease.

Dextran has been used in the past in the critical care setting of human as a volume expander with the rare side effects of anaphylaxis and nephrotoxicity. It has also been used in human coronary arteries with iOCT as a blood displacement medium. Finally it has been used with iOCT in a proximal occlusion model. The main complaint in the final study was a burning sensation that lasted < 10s.

Iodinated contrast is the current gold standard for infrainguinal angiography imaging in patients without renal insufficiency and has also been used with iOCT to improve image quality in human coronary arteries as well as carotid arteries. The current debate in the literature for iOCT medium is between iodinated contrast and dextran and CO2 may offer a superior method of iOCT imaging during lower extremity occlusive disease interventions.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* English speaking
* Scheduled to undergo an infrainguinal angiogram and/or endovascular procedure as determined by a vascular surgery specialist
* Superficial Femoral Artery diseased segment

Exclusion Criteria:

* Acute or Chronic Renal insufficiency with Cr >1.5
* Chronic obstructive pulmonary disease
* Congestive heart failure (American Heart Association C lass III or IV)
* Acute limb ischemia, defined by a significant change in symptoms (one category on the Rutherford scale within the previous 14 days)
* Concurrent oral anticoagulant therapy that cannot be safely withheld

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vikram S Kashyap, MD, Principal Investigator — UH Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Hirsch AT, Criqui MH, Treat-Jacobson D, Regensteiner JG, Creager MA, Olin JW, Krook SH, Hunninghake DB, Comerota AJ, Walsh ME, McDermott MM, Hiatt WR. Peripheral arterial disease detection, awareness, and treatment in primary care. JAMA. 2001 Sep 19;286(11):1317-24. doi: 10.1001/jama.286.11.1317. PMID 11560536
- [Background] Chamie D, Wang Z, Bezerra H, Rollins AM, Costa MA. Optical Coherence Tomography and Fibrous Cap Characterization. Curr Cardiovasc Imaging Rep. 2011 Aug;4(4):276-283. doi: 10.1007/s12410-011-9090-8. Epub 2011 May 12. PMID 21949565
- [Background] Jones MR, Attizzani GF, Given CA 2nd, Brooks WH, Costa MA, Bezerra HG. Intravascular frequency-domain optical coherence tomography assessment of atherosclerosis and stent-vessel interactions in human carotid arteries. AJNR Am J Neuroradiol. 2012 Sep;33(8):1494-501. doi: 10.3174/ajnr.A3016. Epub 2012 Mar 15. PMID 22422179
- [Background] Stefano GT, Mehanna E, Parikh SA. Imaging a spiral dissection of the superficial femoral artery in high resolution with optical coherence tomography-seeing is believing. Catheter Cardiovasc Interv. 2013 Feb;81(3):568-72. doi: 10.1002/ccd.24292. Epub 2012 Apr 17. PMID 22511464
- [Background] Ozaki Y, Kitabata H, Tsujioka H, Hosokawa S, Kashiwagi M, Ishibashi K, Komukai K, Tanimoto T, Ino Y, Takarada S, Kubo T, Kimura K, Tanaka A, Hirata K, Mizukoshi M, Imanishi T, Akasaka T. Comparison of contrast media and low-molecular-weight dextran for frequency-domain optical coherence tomography. Circ J. 2012;76(4):922-7. doi: 10.1253/circj.cj-11-1122. Epub 2012 Feb 3. PMID 22301848
- [Background] Goodney PP, Beck AW, Nagle J, Welch HG, Zwolak RM. National trends in lower extremity bypass surgery, endovascular interventions, and major amputations. J Vasc Surg. 2009 Jul;50(1):54-60. doi: 10.1016/j.jvs.2009.01.035. Epub 2009 May 28. PMID 19481407
- [Background] Li QX, Fu QQ, Shi SW, Wang YF, Xie JJ, Yu X, Cheng X, Liao YH. Relationship between plasma inflammatory markers and plaque fibrous cap thickness determined by intravascular optical coherence tomography. Heart. 2010 Feb;96(3):196-201. doi: 10.1136/hrt.2009.175455. Epub 2009 Oct 28. PMID 19875365
- [Background] Kataiwa H, Tanaka A, Kitabata H, Matsumoto H, Kashiwagi M, Kuroi A, Ikejima H, Tsujioka H, Okochi K, Tanimoto T, Yamano T, Takarada S, Nakamura N, Kubo T, Mizukoshi M, Hirata K, Imanishi T, Akasaka T. Head to head comparison between the conventional balloon occlusion method and the non-occlusion method for optical coherence tomography. Int J Cardiol. 2011 Jan 21;146(2):186-90. doi: 10.1016/j.ijcard.2009.06.059. Epub 2009 Aug 7. PMID 19664829
- [Background] Brezinski M, Saunders K, Jesser C, Li X, Fujimoto J. Index matching to improve optical coherence tomography imaging through blood. Circulation. 2001 Apr 17;103(15):1999-2003. doi: 10.1161/01.cir.103.15.1999. PMID 11306530
- [Background] Xu X, Yu L, Chen Z. Optical clearing of flowing blood using dextrans with spectral domain optical coherence tomography. J Biomed Opt. 2008 Mar-Apr;13(2):021107. doi: 10.1117/1.2909673. PMID 18465956
- [Background] Hoang KC, Edris A, Su J, Mukai DS, Mahon S, Petrov AD, Kern M, Ashan C, Chen Z, Tromberg BJ, Narula J, Brenner M. Use of an oxygen-carrying blood substitute to improve intravascular optical coherence tomography imaging. J Biomed Opt. 2009 May-Jun;14(3):034028. doi: 10.1117/1.3153895. PMID 19566321
- [Background] Hawkins IF, Cho KJ, Caridi JG. Carbon dioxide in angiography to reduce the risk of contrast-induced nephropathy. Radiol Clin North Am. 2009 Sep;47(5):813-25, v-vi. doi: 10.1016/j.rcl.2009.07.002. PMID 19744596
- [Background] Kerns SR, Hawkins IF Jr. Carbon dioxide digital subtraction angiography: expanding applications and technical evolution. AJR Am J Roentgenol. 1995 Mar;164(3):735-41. doi: 10.2214/ajr.164.3.7863904.
- [Background] Moos JM, Ham SW, Han SM, Lew WK, Hua HT, Hood DB, Rowe VL, Weaver FA. Safety of carbon dioxide digital subtraction angiography. Arch Surg. 2011 Dec;146(12):1428-32. doi: 10.1001/archsurg.2011.195. PMID 22288088
- [Background] Weaver FA, Pentecost MJ, Yellin AE, Davis S, Finck E, Teitelbaum G. Clinical applications of carbon dioxide/digital subtraction arteriography. J Vasc Surg. 1991 Feb;13(2):266-72; discussion 272-3. PMID 1899274
- [Background] Hawkins IF, Caridi JG. Carbon dioxide (CO2) digital subtraction angiography: 26-year experience at the University of Florida. Eur Radiol. 1998;8(3):391-402. doi: 10.1007/s003300050400. PMID 9510571
- [Background] Groeneveld AB, Navickis RJ, Wilkes MM. Update on the comparative safety of colloids: a systematic review of clinical studies. Ann Surg. 2011 Mar;253(3):470-83. doi: 10.1097/SLA.0b013e318202ff00. PMID 21217516
- [Background] Kubo T, Nakamura N, Matsuo Y, Okumoto Y, Wu X, Choi SY, Komukai K, Tanimoto T, Ino Y, Kitabata H, Kimura K, Mizukoshi M, Imanishi T, Akagi H, Yamamoto T, Akasaka T. Virtual histology intravascular ultrasound compared with optical coherence tomography for identification of thin-cap fibroatheroma. Int Heart J. 2011;52(3):175-9. doi: 10.1536/ihj.52.175. PMID 21646741
- [Background] Karnabatidis D, Katsanos K, Paraskevopoulos I, Diamantopoulos A, Spiliopoulos S, Siablis D. Frequency-domain intravascular optical coherence tomography of the femoropopliteal artery. Cardiovasc Intervent Radiol. 2011 Dec;34(6):1172-81. doi: 10.1007/s00270-010-0092-8. Epub 2010 Dec 30. PMID 21191586
- [Derived] Kendrick DE, Allemang MT, Gosling AF, Nagavalli A, Kim AH, Nishino S, Parikh SA, Bezerra HG, Kashyap VS. Dextran or Saline Can Replace Contrast for Intravascular Optical Coherence Tomography in Lower Extremity Arteries. J Endovasc Ther. 2016 Oct;23(5):723-30. doi: 10.1177/1526602816657392. Epub 2016 Jul 5. PMID 27385151
- See also: Harrington Heart and Vascular Institute — http://www.uhhospitals.org/services/heart-and-vascular/institute

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were eligible for the study if they were undergoing elective diagnostic angiography for femoropopliteal occlusive disease as indicated by preoperative segmental pressure recordings in an accredited vascular laboratory.
Period: Overall Study
Arm/Group | iOCT
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | iOCT
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 23
Diabetes [Count of Participants; unit: Participants] | 13
Smoking History (>20 Years) [Count of Participants; unit: Participants] | 20
Hyperlipidemia [Count of Participants; unit: Participants] | 18
Rutherford Category 1-3 [Count of Participants; unit: Participants] — Rutherford Category 1-3 are patients with lifestyle-limiting claudication. These patients have less severe disease than critical limb ischemia (Rutherford 4-5).
  Only 22 participants were categorized for this measure.
  Participants | 9
Rutherford Category 4-5 [Count of Participants; unit: Participants] — Rutherford Category 4-5 are patients with critical limb ischemia. These patients have more severe disease than lifestyle-limiting claudication (Rutherford 1-3).
  Only 22 participants were categorized for this measure.
  Participants | 13
Pre-Intervention Serum Creatinine [Mean (Standard Deviation); unit: mg/dL] | 1.03 (0.25)
Heart Rate [Mean (Standard Deviation); unit: beats/min] | 68 (12)
Blood Pressure [Mean (Standard Deviation); unit: mm Hg]
  Systolic BP | 140 (24)
  Diastolic BP | 70 (11)
Lumen Diameter [Mean (Standard Deviation); unit: mm] — Lumen diameter at baseline
  mm | 3.99 (0.99)
Rutherford Class Unknown [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Quality of Images
Description: The metric of image quality was the clear imaging field (CIF), which was defined as a cross section in which ≥270° of the vessel wall architecture was visualized. This has been used previously to quantify adequacy of clearance in OCT image comparison. Two independent observers, blinded to the flush medium used, analyzed all OCT frames in each pullback sequence. Any disagreement >10% was resolved with a consensus re-evaluation at a later time point by the same reviewers. Each individual cross section was assigned a designation of quality or insufficient quality; thus, a quality image proportion was generated for each run by taking the mean of each observer's determinations
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: Clear imaging field (CIF) proportion
Groups:
- Heparinized Saline: Media #4: Heparinized Normal Saline (Heparin NS) will be hand injected using 20 mL (2 U/mL) in antegrade fashion.
Arm/Group | Contrast Injection | Dextran Injection | CO2 Injection | Heparinized Saline
Number analyzed (Participants) | 19 | 19 | 19 | 19
Clear imaging field (CIF) proportion | .702 (.305) | .872 (.12) | .10 (.104) | .743 (.248)

2. Secondary Outcome: Superficial Femoral Artery Plaque Composition by Flush Medium
Time Frame: 1 month
Measure: Number; unit: percentage of plaque composition
Groups:
- Overall: Overall percentage of plaque morphology characterization
Arm/Group | Contrast Injection | Dextran Injection | Heparinized Saline | Overall
Number analyzed (Participants) | 19 | 19 | 19 | 19
percentage of plaque composition
  Fibrotic, % | 57.9 | 62.1 | 63.0 | 61.0
  Calcific, % | 6.9 | 5.5 | 5.4 | 6.0
  Lipid, % | 9.1 | 6.3 | 6.5 | 7.3
  Normal, % | 24.4 | 25.6 | 22.9 | 24.3

ADVERSE EVENTS:
Time Frame: Adverse event data were collected throughout the entire study period. No observed adverse events occurred during the 30-day study period.
Arm/Group | Contrast Injection | Dextran Injection | CO2 Injection | Heparinized Saline
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23 | 0/23 | 0/23

LIMITATIONS AND CAVEATS:
This was a single-center case series that was powered to detect only large differences in image quality. Subtle differences between the 3 liquid media may not have been appreciated despite analysis of over 10,000 individual frames.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No